CLINICAL TRIAL: NCT02110368
Title: An Open-Label, Randomized, Balanced, Single-Dose, Two Treatment, Four Period, Two Sequence Replicate Design, Bioequivalence Study Of Testosterone Topical Gel, 1.62% Metered Pump, Manufactured By Amneal Pharmaceuticals LLC With AndroGel (Testosterone Gel) 1.62% Metered-Dose Pump, Marketed By Abbvie Inc., In Testosterone-Deficient (Hypogonadal) Adult Male Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Test and Reference Testosterone Topical Gel, 1.62% Metered Pump in Testosterone Deficient Adult Male Subjects Under Fasting Conditions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amneal Pharmaceuticals, LLC (Industry)
Collaborators: Phase One Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AL1401
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Primary Hypogonadism; Hypogonadotropic Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AndroGel (Active Comparator): AndroGel (testosterone gel) 1.62% Metered-Dose Pump. One actuation 20.25 mg
  Interventions: Drug: AndroGel (testosterone gel) 1.62% Metered-Dose Pump
- Testosterone Gel (Experimental): Testosterone Topical Gel, 1.62% Metered Pump. One actuation of 20.25 mg.
  Interventions: Drug: Testosterone Topical Gel, 1.62% Metered Pump

INTERVENTIONS:
Drug: Testosterone Topical Gel, 1.62% Metered Pump
  Arms: Testosterone Gel
Drug: AndroGel (testosterone gel) 1.62% Metered-Dose Pump
  Arms: AndroGel

SUMMARY:
Bioequivalence study comparing the rate and extent of testosterone absorption for a test formulation versus the reference product.

DETAILED DESCRIPTION:
To compare the rate and extent of testosterone absorption for a test formulation of Testosterone Topical Gel, 1.62% Metered Pump, manufactured with that of AndroGel® (testosterone gel) 1.62% Metered-Dose Pump, in normal, healthy, adult, testosterone-deficient (hypogonadal) human male subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men with hypogonadism with testosterone levels <250ng/dL
* 18 to 65 years of age (inclusive)
* Have normal PSA < 4.0ng/mL
* Weighing a minimum of 50 kg and having a body mass index between 18.0 and 38.0 kg/m2.
* Good health as determined by medical history and lack of clinically significant abnormalities (other than hypogonadism).
* Vital signs, must be within the following ranges heart rate: 45-100 bpm; systolic BP: 90-150 mmHg; diastolic BP: 50-90 mmHg. Out-of-range vital signs may be repeated.

Exclusion Criteria:

* Is female
* History of allergy or sensitivity to AndroGel® or any component of drug or a related testosterone drug, Axiron®, Testim®, etc.
* History of allergy or intolerance to soy, soybean, and/or soy lecithin
* History of any drug or food hypersensitivity or intolerance which, would compromise the safety of the subject or the study.
* History or presence of clinically significant ocular, cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any othercondition that, would jeopardize the safety of the subject or the validity of the study results.
* Had no major surgery or illness within 3 months before screening.
* History or presence of benign prostate hypertrophy, prostate and/or breast cancer.
* Has tattooed, damaged, scarred skin or any skin condition on right or left upper arm and shoulder region that may affect absorption of drug.
* Has a clinically significant abnormal finding on the physical exam, medical history, electrocardiogram or clinical laboratory results at screening.
* Has been on a significantly abnormal diet during the 4 weeks preceding the first dose of study medication.
* Has donated blood within 56 days or plasma within 30 days prior to the first dose of study medication.
* Has participated in another clinical trial within 30 days prior to the first dose of study medication.
* Has used any over-the-counter medication, including nutritional supplements, within 7 days prior to the first dose of study medication.
* Has used any prescription medication including hormonal treatment and or supplement within 30 days prior to the first dose of study medication.
* No depot injections or drug implants within 3 months of first dose of study medication.
* Has been treated with any known drugs that are moderate or strong inhibitors/inducers of CYP enzymes such as barbiturates, phenothiazine, cimetidine, carbamazepine, etc., within 30 days prior to the first dose of study medication and that may impact subject safety or the validity of the study results.
* Has positive cotinine test and/or smoked or used tobacco products within 60 days prior to the first dose of study medication
* Has a positive urine screen for drugs of abuse
* Has positive alcohol breathalyzer test
* Has a positive test for Hepatitis B surface antigen, Hepatitis C antibody, or Human Immunodeficiency Virus (HIV) at screening or has been previously treated for Hepatitis B, Hepatitis C, or HIV infection.
* Any difficulty fasting or has any dietary restrictions such as lactose intolerance, vegan, low-fat, etc.
* Unavailable for any confinement days or scheduled visits.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-03; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
AUC0-t | Pre-Deose: -1 hour, -0.5 hour and Post-Dose 1, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 32, 36, 40, 48, and 60 hours
  Area under the concentration vs. time curve, from the time of first dosing to the time of the last measured concentration.
AUC0-inf | Pre-Deose: -1 hour, -0.5 hour and Post-Dose 1, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 32, 36, 40, 48, and 60 hours
  Area under the concentration vs. time curve, from time of first dosing to infinity
Cmax | Pre-Deose: -1 hour, -0.5 hour and Post-Dose 1, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 32, 36, 40, 48, and 60 hours
  Maximum reported concentration. Estimated for both baseline

SECONDARY OUTCOMES:
Tmax | Pre-Deose: -1 hour, -0.5 hour and Post-Dose 1, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 32, 36, 40, 48, and 60 hours
  Time at which Cmax is first observed
Kel | Pre-Deose: -1 hour, -0.5 hour and Post-Dose 1, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 32, 36, 40, 48, and 60 hours
  Apparent first order terminal elimination rate constant determined from the terminal log-linear concentration-time data
T 1/2 | Pre-Deose: -1 hour, -0.5 hour and Post-Dose 1, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 32, 36, 40, 48, and 60 hours
  Terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Galitz, MD, Principal Investigator — Phae 1 Solutions
Locations (1):
- Phase One Solutions, Inc., Miami Gardens, Florida, United States